CLINICAL TRIAL: NCT06157333
Title: Effect of Accelerated Repetitive Transcranial Magnetic Stimulation on Depression Symptoms in Patients With Subacute Ischemic Stroke
Brief Title: Efficacy of Accelerated Repetitive Transcranial Magnetic Stimulation on Patients With Post-stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hande Yakar, medical doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-Dryakar
Record Dates: First submitted 2023-11-24; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Post-stroke Depression
Keywords: Accelerated rTMS; Repetitive Transcranial Magnetic Stimulation; Post-stroke Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS group (Active Comparator): We determined the motor threshold (MT) of the contralateral abductor pollicis brevis muscle as the target muscle by stimulating the left motor cortex. The MT was defined as the stimulus intensity required to produce motor evoked potentials of> 50 mV peak-to-peak amplitude in five out of ten consecutive trials in the right abductor pollicis brevis. The rTMS was performed over the left F3 on the scalp according to the 10/20 electroencephalography system with an 8-shaped 70-mm coil. The protocol included high frequency (10 Hz) rTMS applied over the left DLPFC at 110% RMT for two sessions per day, over two weeks for a total of 20 sessions. In each session, a total of 2000 pulses were stimulated for 5 seconds, applied at 25-second intervals, and each rTMS session lasted 20 minutes. Patients were given the opportunity to rest for 1-3 hours in between sessions. A total of 4000 pulses were applied to the patients in one day.
  Interventions: Device: The Magstim Rapid2 Plus Magnetic Stimulator (Magstim, Whitland, Dyfed, UK)
- Sham group (Placebo Comparator): Similar protocol was applied and sham rTMS treatment was given with a sham coil to the sham group.
  Interventions: Device: The Magstim Rapid2 Plus Magnetic Stimulator (Magstim, Whitland, Dyfed, UK)

INTERVENTIONS:
Device: The Magstim Rapid2 Plus Magnetic Stimulator (Magstim, Whitland, Dyfed, UK) — The Magstim Rapid2 Plus Magnetic Stimulator (Magstim, Whitland, Dyfed, UK) device available in our center was used.

SUMMARY:
The FDA approved repetitive transcranial magnetic stimulation (rTMS) for patients with Major Depressive Disorder (MDD) in 2008. The conventional rTMS protocol that has been used effectively for major depression is 5 days per week for 4-6 weeks. The accelerated rTMS protocol involves conducting more than one session per day. In the treatment of post-stroke depression (PSD); although the effectiveness of conventional rTMS procedure has been shown in many studies, there is limited data on accelerated rTMS protocol in which the number of daily sessions is increased. In this study, we aimed to evaluate the efficacy of accelerated rTMS treatment on depression symptoms in patients diagnosed with PSD and whose depressive symptoms persist despite medical treatment, by comparing it with sham stimulation.

Question 1: Is accelerated rTMS an effective and reliable method in the treatment of post-stroke depression? Question 2: Is accelerated rTMS effective on quality of life, functional assessment and motor recovery in patients with post-stroke depression?

DETAILED DESCRIPTION:
Objective: Depression is a complication that negatively affects the quality of life and functional recovery of stroke patients and is associated with increased physical disability, cognitive and social impairment. In addition to being resistant to pharmacotherapy, the side-effect profile of the drugs used in the treatment and the increase in stroke recurrence, increase the need for new alternatives in the treatment of post-stroke depression (PSD). Repetitive transcranial magnetic stimulation (rTMS) is one of the treatment of interest in this field. In the treatment of PSD; although the effectiveness of conventional rTMS procedure has been shown in many studies, there is limited data on accelerated rTMS protocol in which the number of daily sessions is increased. In this study, we aimed to evaluate the efficacy of accelerated rTMS treatment on depression symptoms in patients diagnosed with PSD and whose depressive symptoms persist despite medical treatment, by comparing it with sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke in only one hemisphere is diagnosed by MRI,
* Ischemic stroke within 1-6 months,
* Diagnosis of major depression according to DSM-5 diagnostic criteria by a psychiatrist during post-stroke evaluations,
* Hamilton Depression Rating Scale (HAMD) score of ≥8 as assessed by a clinical psychologist, despite receiving at least one antidepressant treatment,
* Drug use should be stable for at least 2 weeks before accelerated rTMS treatment for depression treatment and no change in drug dose should be made for 6 weeks following treatment,
* Mini mental test score ≥ 24

Exclusion Criteria:

* Known history of epilepsy, dementia, cognitive impairment, neurodegenerative disease,
* İntracranial metallic implant (cochlear implant, brain pacemaker, drug pump, etc.),
* Lesions in the brain due to vascular, traumatic, tumoral or infectious reasons,
* Recurrent strokes,
* Aphasia,
* Alcoholism,
* Pregnancy,
* Cardiac pacemaker,
* Patients diagnosed with psychiatric diseases other than depression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) | The depression severity of the patients was recorded by the clinical psychologist before the treatment, at the end of the treatment and 4 weeks after the end of the treatment.
  The HAMD is the most widely used clinician-administered depression assessment scale. The original version contains 17 items pertaining to symptoms of depression experienced over the past week. By adding up the ratings, 0-53 points are obtained. 0-7 points indicate no depression, 8-15 points indicate mild depression, 16-28 indicates moderate depression, and 29 and above indicates severe depression. The version consisting of 17 items was used in our study, and the patients' response to treatment was evaluated based on these scale scores. At the end of the 2-week rTMS application period; A HAMD score of '7' or below is considered 'Remission', a 50% or more decrease in the HAMD score is considered 'There is a response to treatment', and a decrease of less than 50% in the HAMD score is considered 'No response to treatment'.

SECONDARY OUTCOMES:
Stroke Impact Scale 3.0 (SIS) | Stroke Impact Scale 3.0 was evaluated by the experimenter applying rTMS before the treatment, at the end of treatment and 4 weeks after the end of treatment.
  It is a scale that evaluates the quality of life in hemiplegic patients and consists of 8 subsections (strength, hand function, mobility, communication, activities of daily living, participation, emotion and memory) and 59 questions. The patient is asked to answer each question on a 5-point Likert scale, considering the last week. A score of 1 indicates that the patient could not complete the item, and a score of 5 indicates that the patient completed the item without any difficulty. While evaluating, strength (4-20), thinking-memory (7-35), mood-emotion (9-45), communication (7-35), activities of daily living (10-50), mobility (9-45). Scoring is done separately for 8 subsections: hand function (5-25), participation (8-40). Total score is between 59-295. A low score indicates low quality of life. In addition to 8 subsections, there is a visual analog scale that evaluates the perception of recovery after stroke with a score of 0-100 (0: No recovery, 100: Complete recovery).
Brunnstrom Stages | Brunnstrom Stages was evaluated by the experimenter applying rTMS before treatment, at the end of treatment and 4 weeks after the end of treatment.
  It is a test used to follow motor recovery after stroke. Movement patterns of hemiplegic patients are graded between 1-6.
Functional Independence Measure (FIM) | Functional Independence Measure was evaluated by the experimenter applying rTMS before treatment, at the end of treatment and 4 weeks after the end of treatment.
  The general body functions of the individual are evaluated with 6 sub-main sections under the headings of four motor (self-care, sphincter control, transfer and displacement) and two cognitive activities (communication and social cognition). Each subsection contains articles in its own category. Motor functions are evaluated in 13 items and cognitive functions in 5 items, and the scale consists of a total of 18 items. Each item is scored using a 7-point Likert scale, with the highest score being 7 and the lowest score being 1, depending on the patient's level of independence in relation to the relevant activity. 1-2 points are considered dependent, 3-5 points are considered partially dependent, and 6-7 points are considered independent. By summing the scores of 18 items, a total score between 18-126 is obtained. A score of 18 points indicates that the individual is completely dependent, while a score of 126 indicates complete independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen X, Liu M, Cheng Y, Jia C, Pan X, Gou Q, Liu X, Cao H, Zhang L. Repetitive transcranial magnetic stimulation for the treatment of post-stroke depression: A systematic review and meta-analysis of randomized controlled clinical trials. J Affect Disord. 2017 Mar 15;211:65-74. doi: 10.1016/j.jad.2016.12.058. Epub 2017 Jan 10. PMID 28092847
- [Background] Gaynes BN, Lux L, Gartlehner G, Asher G, Forman-Hoffman V, Green J, Boland E, Weber RP, Randolph C, Bann C, Coker-Schwimmer E, Viswanathan M, Lohr KN. Defining treatment-resistant depression. Depress Anxiety. 2020 Feb;37(2):134-145. doi: 10.1002/da.22968. Epub 2019 Oct 22. PMID 31638723
- [Background] Klomjai W, Katz R, Lackmy-Vallee A. Basic principles of transcranial magnetic stimulation (TMS) and repetitive TMS (rTMS). Ann Phys Rehabil Med. 2015 Sep;58(4):208-213. doi: 10.1016/j.rehab.2015.05.005. Epub 2015 Aug 28. PMID 26319963
- [Background] Horvath JC, Mathews J, Demitrack MA, Pascual-Leone A. The NeuroStar TMS device: conducting the FDA approved protocol for treatment of depression. J Vis Exp. 2010 Nov 12;(45):2345. doi: 10.3791/2345. PMID 21189465
- [Background] Liu C, Wang M, Liang X, Xue J, Zhang G. Efficacy and Safety of High-Frequency Repetitive Transcranial Magnetic Stimulation for Poststroke Depression: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2019 Oct;100(10):1964-1975. doi: 10.1016/j.apmr.2019.03.012. Epub 2019 Apr 17. PMID 31002813
- [Background] Shao D, Zhao ZN, Zhang YQ, Zhou XY, Zhao LB, Dong M, Xu FH, Xiang YJ, Luo HY. Efficacy of repetitive transcranial magnetic stimulation for post-stroke depression: a systematic review and meta-analysis of randomized clinical trials. Braz J Med Biol Res. 2021 Jan 15;54(3):e10010. doi: 10.1590/1414-431X202010010. eCollection 2021. PMID 33470386
- [Background] Frey J, Najib U, Lilly C, Adcock A. Novel TMS for Stroke and Depression (NoTSAD): Accelerated Repetitive Transcranial Magnetic Stimulation as a Safe and Effective Treatment for Post-stroke Depression. Front Neurol. 2020 Aug 11;11:788. doi: 10.3389/fneur.2020.00788. eCollection 2020. PMID 32849235
- [Background] Williams JB. A structured interview guide for the Hamilton Depression Rating Scale. Arch Gen Psychiatry. 1988 Aug;45(8):742-7. doi: 10.1001/archpsyc.1988.01800320058007. PMID 3395203
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Frank E, Prien RF, Jarrett RB, Keller MB, Kupfer DJ, Lavori PW, Rush AJ, Weissman MM. Conceptualization and rationale for consensus definitions of terms in major depressive disorder. Remission, recovery, relapse, and recurrence. Arch Gen Psychiatry. 1991 Sep;48(9):851-5. doi: 10.1001/archpsyc.1991.01810330075011. PMID 1929776
- [Background] Kucukdeveci AA, Yavuzer G, Tennant A, Suldur N, Sonel B, Arasil T. Adaptation of the modified Barthel Index for use in physical medicine and rehabilitation in Turkey. Scand J Rehabil Med. 2000 Jun;32(2):87-92. PMID 10853723
- [Background] Lai SM, Studenski S, Duncan PW, Perera S. Persisting consequences of stroke measured by the Stroke Impact Scale. Stroke. 2002 Jul;33(7):1840-4. doi: 10.1161/01.str.0000019289.15440.f2. PMID 12105363